CLINICAL TRIAL: NCT02446847
Title: A Phase 2, Open Label Study of the Safety, Antiretroviral Activity and Pharmacokinetics of 3BNC117 During a Short Analytical Treatment Interruption in HIV-infected Subjects
Brief Title: 3BNC117 Monoclonal Antibody in HIV-infected Subjects During Treatment Interruption
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCA-0867
Record Dates: First submitted 2015-03-17; First posted 2015-05-18 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: HIV-1 Infection
Keywords: HIV; 3BNC117; Broadly neutralizing antibody
MeSH Terms: interventions — 3BNC117 antibody; Treatment Interruption

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: 3BNC117 IV + ART Interruption (Experimental): Two intravenous infusions of 3BNC117 (30 mg/kg) at day 0 and day 21, with interruption of antiretroviral treatment (ART) at day 2.
  Interventions: Drug: 3BNC117; Other: ART Interruption
- Group B: 3BNC117 IV + ART interruption (Experimental): Four intravenous infusions of 3BNC117 (30 mg/kg) at day 0, day 14, day 28, and day 42 with interruption of antiretroviral treatment (ART) at day 2.
  Interventions: Drug: 3BNC117; Other: ART Interruption

INTERVENTIONS:
Drug: 3BNC117 — 3BNC117 infusions
  Other Names: 3BNC117 antibody
Other: ART Interruption — Antiretroviral therapy will be discontinued 2 days after the first 3BNC117 infusion (day 2) and resumed at week 12.
  Other Names: Treatment Interruption

SUMMARY:
This study evaluates the effects of two infusions of 3BNC117 in preventing or delaying rebound of viral load during a brief treatment interruption of standard ART and its safety during a brief analytical interruption of antiretroviral therapy.

DETAILED DESCRIPTION:
The proposed study is a Phase II, open label study to evaluate the safety and antiretroviral activity of two and four infusions of 3BNC117 in HIV-infected subjects on combination ART during a brief analytical treatment interruption.

After meeting enrollment criteria sixteen subjects with 3BNC117 sensitive virus (<2μg/ml IC50) will receive two (Group A) or four (Group B) intravenous infusions of 3BNC117, administered at 30 mg/kg.

In both dosing groups, antiretroviral therapy will be discontinued 2 days after the first 3BNC117 infusion (day 2) until week 12. Combination ART will be resumed at week 12. ART will be resumed sooner if plasma HIV-1 RNA level is ≥ 200 copies/ml or if CD4+ count drops < 350 cells/μl and either result is confirmed upon repeat measurement. Participants will be followed weekly until week 12 for safety assessments and for monitoring plasma HIV-1 RNA levels (viral load). CD4+ T cell counts will be monitored every 2 weeks until week 12.

Participants may remain off antiretroviral therapy after week 12, with weekly viral load monitoring, if viral rebound does not occur by week 12. Participants will be followed for a total of 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* HIV-1 infection confirmed by ELISA and immunoblot.
* Plasma HIV-1 RNA < 50 copies/ml for at least 12 months while on combination ART and < 20 copies/ml at the screening visit. [Note: One or two viral blips of < 200 copies/mL prior to enrollment are permitted if preceded and followed by test results showing VL less than or equal to 50 copies/mL on the same ARV regimen.]
* 3BNC117 sensitivity (IC50 < 2 μg/ml) of subject derived HIV-1 virus isolates. These are isolated under protocol MCA-823 by co-culture of subject PBMCs with HIV-uninfected donor PBMCs followed by in vitro neutralization assays as previously described
* Current CD4 cell count > 500 cells/μl and no prior CD4 cell count < 200 cells/μl.
* Willing to interrupt antiretroviral treatment for 12 weeks, or until viral rebound occurs.
* If sexually active male or female, and participating in sexual activity that could lead to pregnancy using an effective method of contraception throughout the study period. Subjects should also agree to use a male or female condom during the time of pausing their HIV medication.
* If on an NNRTI-based regimen willing to a switch for 4 weeks to dolutegravir.

Exclusion Criteria:

* Have a history of AIDS-defining illness within 1 year prior to enrollment
* History of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the trial physician within the last 6 months;
* Chronic hepatitis B or hepatitis C;
* Patient report, or chart history, of significant coronary artery disease, myocardial infarction, percutaneous coronary intervention with placement of cardiac stents;
* Patient report, or chart history, of diabetes type 1 or 2 and/or current use of insulin or oral hypoglycemic medications;
* Uncontrolled hypertension, as defined by a systolic blood pressure > 180 and/or diastolic blood pressure > 120, in the presence or absence of anti-hypertensive medications;
* Any other clinically significant acute or chronic medical condition, such as autoimmune diseases, that in the opinion of the investigator would preclude participation;
* Current cigarette use in excess of 1 pack per day;
* Laboratory abnormalities in the parameters listed below:

  * Absolute neutrophil count ≤1,000
  * Hemoglobin ≤ 10 gm/dL
  * Platelet count ≤125,000
  * ALT ≥ 2.0 x ULN
  * AST ≥ 2.0 x ULN
  * Total bilirubin ≥ 1.5 ULN
  * Creatinine ≥ 1.1 x ULN
  * Coagulation parameters ≥ 1.5 x ULN;
* Current antiretroviral regimen includes either maraviroc or enfuvirtide;
* Pregnancy or lactation;
* Any vaccination within 14 days prior to 3BNC117 administration;
* Receipt of any monoclonal antibody therapy of any kind in the past;
* Participation in another clinical study of an investigational product currently or within past 12 weeks, or expected participation during this study.
* History of resistance to two or more antiretroviral drug classes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2017-03-25 (Actual); Study Completion 2017-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, MD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A: 3BNC117 IV + ART Interruption | Group B: 3BNC117 IV + ART Interruption
Started | 8 | 8
Completed | 8 | 6
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: 3BNC117 IV + ART Interruption | Group B: 3BNC117 IV + ART Interruption | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Full Range); unit: years] | 46 [26 to 62] | 38 [27 to 59] | 42 [26 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 5 | 8
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Virologic Rebound at 8 Weeks After Interruption of Antiretroviral Therapy
Description: Virologic rebound is defined as confirmed plasma HIV-1 RNA level > 200 copies/ml in two separate occasions
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 3BNC117 IV + ART Interruption | Group B: 3BNC117 IV + ART Interruption
Number analyzed (Participants) | 6 | 8
Participants | 4 | 3

2. Primary Outcome: The Rate of Signs, Symptoms and Laboratory Abnormalities After 3BNC117 Infusions
Description: The percentage of participants who experienced adverse events (e.g. signs, symptoms and laboratory abnormalities) following 3BNC117 infusions.
Time Frame: 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 3BNC117 IV + ART Interruption | Group B: 3BNC117 IV + ART Interruption
Number analyzed (Participants) | 8 | 8
Participants | 8 | 8

3. Secondary Outcome: The Plasma Level of 3BNC117 at the Time of Viral Rebound.
Description: The plasma concentrations of 3BNC117 at the time of viral rebound (i.e. confirmed plasma HIV-1 RNA levels > 200 copies/ml).
Time Frame: 36 weeks
Population: Two participants excluded from analysis because of detectable plasma HIV-1 RNA levels prior to first administration of the investigational product.
Measure: Mean (Standard Deviation); unit: micrograms/ml
Arm/Group | Group A: 3BNC117 IV + ART Interruption | Group B: 3BNC117 IV + ART Interruption
Number analyzed (Participants) | 6 | 7
micrograms/ml | 61.15 (42.41) | 74.37 (65.17)

ADVERSE EVENTS:
Time Frame: Participants were followed for 36 weeks from enrollment.
Arm/Group | Group A: 3BNC117 IV + ART Interruption | Group B: 3BNC117 IV + ART Interruption
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/8
Other Adverse Events (participants affected / at risk) | 6/8 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: 3BNC117 IV + ART Interruption (N=8) | Group B: 3BNC117 IV + ART Interruption (N=8)
Transient ischemic attack (Nervous system disorders) | 0 | 1 — The participant was admitted to the hospital with a transient ischemic attach 30 wks after last study intervention. The event was considered not related to the study, but secondary to underlying risk factors.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: 3BNC117 IV + ART Interruption (N=8) | Group B: 3BNC117 IV + ART Interruption (N=8)
Headache (Nervous system disorders) | 6 (7) | 2 (2)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (7)
Paresthesia upper extremity (Nervous system disorders) | 3 (3) | 0 (0)
Chest tightness (Cardiac disorders) | 2 (2) | 0 (0)
Back pain (General disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hyperbilirubinemia (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2015-09-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT02446847/Prot_000.pdf
  • Statistical Analysis Plan (2015-09-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT02446847/SAP_001.pdf
  • Informed Consent Form (2015-09-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT02446847/ICF_002.pdf